CLINICAL TRIAL: NCT06815484
Title: Single-centre, Randomised, Controlled Study Designed to Evaluate the Impact of a Nine-week Supervised Physical Activity Programme Physical Activity Programme on Reducing the Risk of Burnout in Burnout in Carers
Brief Title: Preventing Burnout Among Caregivers Through Physical Activity
Acronym: PACA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-A02575-42
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Burn Out
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Pilot, prospective, comparative, randomised (2 arms), controlled study
Who Masked: Participant, Investigator
Masking Description: The choice of randomisation by minimisation allows participants to be allocated at random to the two groups (intervention and control groups), thus ensuring a balance in the known characteristics likely to influence the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group : adaptive physical activity programme (Experimental): Participants will benefit from an adaptive physical activity programme supervised by a physical activity professional over a 9-week period. Participants will also receive the World Health Organisation's recommendations on physical activity, which recommend at least 150 minutes a week of moderate-intensity activity or 75 minutes of high-intensity activity, and highlight the importance of limiting sedentary behaviour.
  Interventions: Other: Intervention group with physical activity programme; Other: Recommendations of the World Health Organisation
- Control Group : recommendations on physical activity (Active Comparator): Participants will be given only the World Health Organisation's recommendations on physical activity. At the end of the 9-week intervention period, participants will have the opportunity to take part in a motivational interview with a physical activity professional to encourage regular physical activity.
  Interventions: Other: Recommendations of the World Health Organisation

INTERVENTIONS:
Other: Intervention group with physical activity programme — Programme comprising active breaks to be incorporated into daily life, supervised group physical activity sessions with personalised advice and a motivational interview with a physical activity professional to encourage regular physical activity.
  Arms: Intervention group : adaptive physical activity programme
Other: Recommendations of the World Health Organisation — The World Health Organisation's recommendations on physical activity, which recommend at least 150 minutes a week of moderate-intensity activity or 75 minutes of high-intensity activity, and highlight the importance of limiting sedentary behaviour.

SUMMARY:
The purpose of this study is to evaluate the impact of an adaptive physical activity programme to prevent the risk of burnout at the end of the programme (10 weeks after the start of the intervention).

DETAILED DESCRIPTION:
The PACA trial is a pilot, prospective, comparative, randomised (2 arms), controlled, single-centre study.

The study population consisted of adult healthcare professionals at the Clinique de la Sauvegarde with a low to moderate level of physical activity and no contraindications to physical activity.

Participants will be randomised into two arms (ratio 1:1):

* Arm A (intervention): Participants will benefit from an adaptive physical activity programme supervised by a physical activity professional over a 9-week period.
* Arm B (control): Participants will receive the recommendations of the world health organisation for physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years ;
* Non-physician health professionals at the Clinique de la Sauvegarde ;
* Low or moderate level of physical activity, as assessed by the questionnaire International Physical Activity Questionnaire. In fact, work-related physical activity is not associated with a reduction in burnout ;
* Absence of serious chronic pathology incompatible with the physical activity of the protocol ;
* Willing and available to commit to the project for the duration of the study ;
* Using a personal smartphone or tablet and with an Internet connection ;
* Able to read, write and understand French ;
* Membership of a social security scheme.

Exclusion Criteria:

* High level of physical activity (not including work-related physical activity) ;
* Contraindication to physical activity (uncontrolled hypertension, uncontrolled heart disease...) ;
* Concurrent participation in another physical activity study ;
* Pregnant or likely to be pregnant ;
* Unable to be monitored for medical, social, family, geographical or psychological reasons for the duration of the study ;
* Persons deprived of their liberty by judicial or adm inistrative decision, or adults protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Shirom - Melamed Burnout Measure | 10 weeks
  The primary endpoint is the burnout will be measured by the score on the Shirom - Melamed Burnout Measure questionnaire.
  The validated French version of the Shirom-Melamed Burnout Measure comprises 14 items assessed on a Likert scale from 1 (never) to 7 (always), quantifying the frequency of symptoms experienced over the last seven days.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France